CLINICAL TRIAL: NCT02593435
Title: The Registration Program of BRCA1/2 Gene in Chinese Breast Cancer Group
Brief Title: The Registration Program of BRCA1/2 Gene
Acronym: RCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Anti-Cancer Association (Other)
Responsible Party: Sponsor
Other Study IDs: CBRCA
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: BRCA1/2 gene mutation; Breast Cancer; Chinese high risk group
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — The samples, both tissue(s) and blood of patients should be provided for NGS test after ICF being signed
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: There will be two groups, one is breast cancer patient group, another group inlude the first-degree relatives and second degree relatives of patients with BRCA1/2 mutation. All volunteers should provid tissue(s) and blood for NGS test.
  Interventions: Genetic: NGS test

INTERVENTIONS:
Genetic: NGS test — To record the characteristic QC parameters and evaluate the detection performance of Next-Generation Sequencing (NGS), including coverage depth and sequence similarity, then be used to evaluate the quality of base recognition and alignment.
  To know mutation characteristic spectrum of BRCA1/2.

SUMMARY:
Purpose:

1. Screening of large samples is to search the gene mutation of the breast cancer susceptibility gene (BRCA1 and BRCA2) in Chinese high risk group.
2. To build the breast cancer BRCA1/2 mutation database of Chinese group.
3. To build the hazard model of breast cancer BRCA1/2 mutation of Chinese group.

DETAILED DESCRIPTION:
It is the first large-scale and systematic study that fully recognize and review on the mutation spectrum of BRCA1/2 and the risk of Breast cancer in Chinese high risk group, it will be a Landmark research of susceptibility genes in Chinese breast cancer.

ELIGIBILITY:
Chinese Genetic/Familial breast cancer patients, and its first or second degree relatives with breast cancer (female or male).

The selection will be based on NCCN Clinical Practice Guidelines in Oncology (Genetic/Familial High-Risk Assessment: Breast and Ovarian).

Inclusion Criteria:

Patients: it must be from independent family and meet the one or more of the following conditions.

1. Patients' age at diagnosis: 45 years or younger.
2. Patients' age at diagnosis: 50 years or younger.
3. Breast cancer patients: it must meet the one or more of the following family medical histories.

   3.1 Patients' age at diagnosis: 50 years or younger, and the one or more of the next of Kin has breast cancer.

   3.2 Patients' age at diagnosis: any of age, and the one or more of the next of Kin has breast cancer that its age at diagnosis was 50 years or younger.

   3.3 Patients' age at diagnosis: any of age, and the two or more of the next of Kin have breast cancer that its age at diagnosis was 50 years or younger.

   3.4 Patients' age at diagnosis: any of age, and the one or more of the next of Kin has epithelial ovarian cancer.

   3.5 Patients' age at diagnosis: any of age, and the two or more of the next of Kin have pancreatic cancer and/or prostate cancer (Gleason grading>7, any of age).

   3.6 Patients' age at diagnosis: any of age, and the one or more of the close-male relatives has breast cancer.
4. Triple negative patients' age of onset: 60 years or younger.
5. Patients: male and have breast cancer.

Patients' first or second degree relatives are BRCA1/2 mutation carrier (1-5 people):

First or second degree female adult relatives of patients (age: 18 years or older), it will be selected from the same paternal or maternal side according to the family disease.

First or second degree male relatives of patients have breast cancer.

Exclusion Criteria:

N/A.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Chinese Breast Cancer Patients
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Screening of large samples is to search the gene mutation of the breast cancer susceptibility gene (BRCA1 and BRCA2) in Chinese high risk group. | About 2 years

SECONDARY OUTCOMES:
To build the database of the Chinese breast cancer BRCA1/2 mutation. | About 2 years
To build the hazard model of Chinese breast cancer BRCA1/2 mutation. | About 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ze-Fei Jiang, Doctor, Principal Investigator — 307 Hospital of PLA
Locations (1):
- The 307th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The data-sharing of the volunteers' genetic information need be discussed more.